CLINICAL TRIAL: NCT07285889
Title: The Safety and Efficacy of Gecacitinib (Also Known as Jaktinib) Combined Glucocorticoids as First-line Treatment for Grade II-IV Acute Graft-versus-host Disease.
Brief Title: First-Line Jaktinib for Acute Graft-Versus-Host Disease (aGVHD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yi Luo, Professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJU-GVHD-JAKTINIB1
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Graft Versus Host Disease
Keywords: acute graft-versus-host disease; Jaktinib; hematopoietic stem cell transplantation; gecacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gecacitinib (also known as Jaktinib) group (Experimental): Patients accept Gecacitinib (also known as Jaktinib) combined glucocorticoids treatment
  Interventions: Drug: Gecacitinib (also known as Jaktinib) combined glucocorticoids

INTERVENTIONS:
Drug: Gecacitinib (also known as Jaktinib) combined glucocorticoids — This clinical trial employs a standard 3+3 design to establish the Recommended Phase 2 Dose (RP2D) of gecacitinib (also known as jaktinib) combined with methylprednisolone. The dose escalation begins at 50 mg QD. Based on the safety observed in the initial cohort of three subjects, the dose will either be escalated to 50 mg BID or the cohort will be expanded. The subsequent escalation level is to 150 mg QD. Throughout this phase, the methylprednisolone dose is adjusted per the investigator's assessment. After determining the RP2D, the study advances to an efficacy evaluation stage, where approximately 25 additional subjects are enrolled to receive the combination at the RP2D for a minimum of 28 days. The primary objective of the initial phase is to assess safety and tolerability, while the secondary goal of the expansion is to gather preliminary efficacy data on the combination regimen.
  Other Names: gecacitinib (also known as jaktinib)

SUMMARY:
This study aims to evaluate the optimal dose (Recommended Phase 2 Dose, RP2D), preliminary safety, and efficacy of gecacitinib (also known as jaktinib) in combination with glucocorticoids as first-line therapy for patients with grade II-IV acute graft-versus-host disease (aGVHD) following allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
This study is a single-center, single-arm, prospective interventional trial utilizing a 3+3 dose escalation design to evaluate the safety and efficacy of first-line gecacitinib (also known as jaktinib) in combination with glucocorticoids for the treatment of grades II-IV acute graft-versus-host disease (aGVHD) following allogeneic hematopoietic stem cell transplantation (allo-HSCT).

A total of 35 patients will be enrolled across both the dose exploration phase (using the 3+3 design to determine the Recommended Phase 2 Dose [RP2D]) and the efficacy evaluation phase (where additional patients are treated at the RP2D to further assess efficacy and safety).

The primary objectives include:

1. Determining the RP2D of gecacitinib (also known as jaktinib) in combination with glucocorticoids.
2. Assessing the safety profile (e.g., incidence and severity of adverse events).
3. Evaluating efficacy (e.g., overall response rate at Day 28). Secondary endpoints may include duration of response, survival outcomes, and biomarker analyses.

This design is appropriate for early-phase trials seeking to establish dosing and preliminary activity of a novel combination therapy in a high-risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide signed informed consent and be ≥18 years of age at the time of consent.
2. Recipients of allogeneic hematopoietic stem cell transplantation (allo-HSCT) using bone marrow, peripheral blood stem cells, or umbilical cord blood.
3. Have received systemic glucocorticoid therapy for no more than 2 days prior to enrollment.
4. Demonstrate clear myeloid and platelet engraftment: absolute neutrophil count (ANC) > 1.0 × 10⁹/L and platelet count > 50 × 10⁹/L (permitted use of growth factors or transfusion support).
5. Clinical diagnosis of grade II-IV acute GVHD (aGVHD) per the MAGIC (Mount Sinai Acute GVHD International Consortium) criteria (Appendix 1).
6. ECOG performance status of 0-2.
7. Life expectancy > 4 weeks.
8. Able to swallow tablets.
9. Willing and able to comply with study procedures and follow-up.

Exclusion Criteria:

1. History of ≥2 allo-HSCT procedures.
2. Development of aGVHD following unplanned donor lymphocyte infusion (DLI) for relapse of underlying malignancy. Note: Planned DLI as part of the transplant protocol is permitted.
3. Concurrent treatment with another JAK inhibitor. Note: Patients who previously discontinued JAK inhibitors due to toxicity (not refractory aGVHD) are eligible.
4. Active bleeding.
5. Diagnosed or suspected chronic GVHD.
6. Uncontrolled active infection, defined as sepsis-induced hemodynamic instability or progressive symptoms/signs/imaging findings attributable to infection. Asymptomatic or persistent fever alone is not exclusionary.
7. unresolved toxicity or complications from allo-HSCT (excluding aGVHD).
8. Clinically significant abnormalities that may compromise safety, including: a) Uncontrolled diabetes (fasting glucose >13.9 mmol/L); b) Hypertension unresponsive to ≥2 agents (systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg); c) Peripheral neuropathy ≥Grade 2 (per NCI CTCAE v5.0).
9. Within 6 months prior to screening: NYHA Class III/IV heart failure, unstable angina, myocardial infarction, cerebrovascular accident, or pulmonary embolism.
10. Arrhythmia requiring treatment or QTcB interval >480 ms at screening.
11. Severe renal impairment (serum creatinine >1.5 × ULN) at screening.
12. Pre-transplant history of gastrointestinal ulcers, gastrectomy, or intestinal resection that may impair drug absorption.
13. Major surgery within 4 weeks prior to screening without full recovery.
14. Cholestatic disorders or hepatic sinusoidal obstruction syndrome (SOS/VOD) at screening (defined as persistent hyperbilirubinemia and organ dysfunction unrelated to GVHD).
15. Active uncontrolled viral infections at screening: HBV: HBsAg⁺ with detectable HBV-DNA, or detectable HBV-DNA regardless of HBsAg status; HCV: Anti-HCV antibody⁺ with detectable HCV-RNA.
16. History of active tuberculosis within 6 months prior to screening.
17. Epilepsy or current use of psychotropic/sedative medications.
18. Pregnancy, lactation, or intention to conceive; male patients unwilling to use condoms during treatment and for 2 days after the last dose.
19. Other active malignancies (excluding the transplanted hematologic malignancy) within 5 years.
20. Current use of anticoagulants or antiplatelet agents (except low molecular weight heparin).
21. Any condition that, in the investigator's judgment, may compromise patient safety or protocol compliance.
22. Known hypersensitivity to jaktinib, its analogs, or excipients.
23. Participation in another interventional clinical trial within 4 weeks prior to screening.
24. Investigator determination of unsuitability for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Reactions by Dosage Group in Patients with Grade II-IV Acute GVHD Treated with First-Line Gecacitinib (also known as Jaktinib) and corticosteroids | 28 days
  The primary outcome of this study was the incidence of adverse reactions, stratified by Gecacitinib (also known as Jaktinib) dosage group, in patients diagnosed with grade II-IV acute graft-versus-host disease (GVHD) receiving first-line treatment with Gecacitinib (also known as Jaktinib) in combination with corticosteroids.
The Day 28 Overall Response Rate (ORR) in patients with grade II-IV acute graft-versus-host disease (GVHD) treated with Ggecacitinib (also known as Jaktinib) in combination with corticosteroids as first-line therapy. | 28 days
  The Day 28 Overall Response Rate (ORR) in patients with grade II-IV acute graft-versus-host disease (GVHD) treated with Gecacitinib (also known as Jaktinib) in combination with corticosteroids as first-line therapy.

SECONDARY OUTCOMES:
To determine the Recommended Phase 2 Dose (RP2D) of Jaktinib for the efficacy evaluation phase. | 28 days
  To determine the Recommended Phase 2 Dose (RP2D) of Jaktinib for the efficacy evaluation phase.
Overall Response Rate (ORR) at Weeks 1, 2, 6, 8, 12, and 24 following treatment with Jaktinib in combination with corticosteroids. | Weeks 1, 2, 6, 8, 12, and 24
  Overall Response Rate (ORR) at Weeks 1, 2, 6, 8, 12, and 24 following treatment with Jaktinib in combination with corticosteroids.
Duration of Response (DOR) | 1 year
  Defined as the time from the first achievement of response to disease progression of aGVHD, initiation of alternative systemic therapy, or death from any cause.
180-day cumulative non-relapse mortality (NRM) | 180 days
  Defined as the proportion of subjects who die from causes other than progression or relapse of the underlying hematologic malignancy within 180 days from treatment initiation.
Change in levels of serum biomarkers | Days 7, 14, and 28
  Change in levels of serum biomarkers from baseline to Days 7, 14, and 28 following treatment with Jaktinib in combination with corticosteroids.
1-year GVHD-free, relapse-free survival (GRFS) | 1 year
  Defined as the proportion of subjects who are alive and free from relapse of the underlying malignancy and without active chronic GVHD requiring systemic immunosuppressive therapy at 1 year after treatment initiation.
1-year cumulative incidence of moderate-to-severe chronic graft-versus-host disease (cGVHD). | 1 year
  1-year cumulative incidence of moderate-to-severe chronic graft-versus-host disease (cGVHD).
Immune reconstitution at Weeks 4, 12, and 24 post-transplantation | Weeks 4, 12, and 24 post-transplantation
  Immune reconstitution at Weeks 4, 12, and 24 post-transplantation, as assessed by lymphocyte subset counts (CD3⁺ T cells, CD19⁺ B cells, CD56⁺ NK cells).

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the current study are available from the principal investigator upon reasonable request. Access to the data will be granted following review and approval of a methodologically sound research proposal, in compliance with ethical standards and data protection regulations. Data sharing is subject to the execution of a data use agreement to ensure appropriate use and confidentiality.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years
Access Criteria: Access to the data will be granted following review and approval of a methodologically sound research proposal, in compliance with ethical standards and data protection regulations. Data sharing is subject to the execution of a data use agreement to ensure appropriate use and confidentiality.

REFERENCES:
- [Result] Moiseev IS, Morozova EV, Bykova TA, Paina OV, Smirnova AG, Dotsenko AA, Borzenkova ES, Galimov AN, Gudognikova YV, Ekushov KA, Kozhokar PV, Osipova AA, Pirogova OV, Rudakova TA, Klimova OU, Tcvetkov NY, Kulagin EA, Surkova EA, Lapin SV, Rodionov GG, Moiseev SI, Serov YA, Zubarovskaya LS, Afanasyev BV. Long-term outcomes of ruxolitinib therapy in steroid-refractory graft-versus-host disease in children and adults. Bone Marrow Transplant. 2020 Jul;55(7):1379-1387. doi: 10.1038/s41409-020-0834-4. Epub 2020 Feb 18. PMID 32071418
- [Result] Dignan FL, Clark A, Amrolia P, Cornish J, Jackson G, Mahendra P, Scarisbrick JJ, Taylor PC, Hadzic N, Shaw BE, Potter MN; Haemato-oncology Task Force of British Committee for Standards in Haematology; British Society for Blood and Marrow Transplantation. Diagnosis and management of acute graft-versus-host disease. Br J Haematol. 2012 Jul;158(1):30-45. doi: 10.1111/j.1365-2141.2012.09129.x. Epub 2012 Apr 26. PMID 22533831
- [Result] Zeiser R, von Bubnoff N, Butler J, Mohty M, Niederwieser D, Or R, Szer J, Wagner EM, Zuckerman T, Mahuzier B, Xu J, Wilke C, Gandhi KK, Socie G; REACH2 Trial Group. Ruxolitinib for Glucocorticoid-Refractory Acute Graft-versus-Host Disease. N Engl J Med. 2020 May 7;382(19):1800-1810. doi: 10.1056/NEJMoa1917635. Epub 2020 Apr 22. PMID 32320566
- [Result] Jagasia M, Perales MA, Schroeder MA, Ali H, Shah NN, Chen YB, Fazal S, Dawkins FW, Arbushites MC, Tian C, Connelly-Smith L, Howell MD, Khoury HJ. Ruxolitinib for the treatment of steroid-refractory acute GVHD (REACH1): a multicenter, open-label phase 2 trial. Blood. 2020 May 14;135(20):1739-1749. doi: 10.1182/blood.2020004823. PMID 32160294